CLINICAL TRIAL: NCT01583647
Title: A Single Dose Study to Evaluate the Safety, Tolerability and Pharmacokinetics of ER Niacin/Laropiprant in Adolescents With Heterozygous Familial Hypercholesterolemia
Brief Title: A Study of Extended-release (ER) Niacin/Laropiprant in Adolescents With Heterozygous Familial Hypercholesterolemia (MK-0524A-158)
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: In HPS2-THRIVE, MK-0524A did not meet the primary efficacy objective and there was a significant increase in incidence of some types of non-fatal SAEs.
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0524A-158; 2012-001443-49 (EudraCT Number)
Record Dates: First submitted 2012-04-20; First posted 2012-04-24 (Estimated); Results first posted 2013-12-04 (Estimated); Last update posted 2015-11-03 (Estimated); Status verified 2015-11

CONDITIONS: Hypercholesterolemia, Familial; Heterozygous Familial Hypercholesterolemia
MeSH Terms: conditions — Hyperlipoproteinemia Type II | interventions — Niacin; MK-0524

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- MK-0524A 1 g/20 mg (Panel A) (Experimental): Single oral dose of 1 tablet of MK-0524A. Each tablet contained Extended Release (ER) Niacin 1g and laropiprant 20 mg
  Interventions: Drug: MK-0524A
- MK-0524A 2 g/40 mg (Panel B) (Experimental): Single oral dose of 2 tablets of MK-0524A. Each tablet contained Extended Release (ER) Niacin 1g and laropiprant 20 mg
  Interventions: Drug: MK-0524A

INTERVENTIONS:
Drug: MK-0524A — 1 tablet of MK-0524A (1g ER niacin/20mg laropripant) orally
  Other Names: Extended-release (ER) Niacin/Laropiprant
  Arms: MK-0524A 1 g/20 mg (Panel A)
Drug: MK-0524A — 2 tablets of MK-0524A (1g ER niacin/20mg laropripant) orally
  Other Names: Extended-release (ER) Niacin/Laropiprant
  Arms: MK-0524A 2 g/40 mg (Panel B)

SUMMARY:
The purpose of this study is to determine the pharmacokinetics of laropiprant following administration of a single dose of 1 (Panel A) and 2 (Panel B) combination tablets of MK-0524A in adolescents with heterozygous familial hypercholesterolemia.

ELIGIBILITY:
Inclusion Criteria:

* Post-pubescent adolescent age 10 to 16 with heterozygous familial hypercholesterolemia
* Agree to use (and/or have their partner use) acceptable methods of birth control beginning at the prestudy visit until at least 2 weeks after dosing of study drug
* Height and weight fall between the 10th and 95th percentile for age with a minimum body weight of 23 kg
* Receiving appropriate medical care for hypercholesterolemia, such as a statin or other lipid-modifying therapy.

Exclusion Criteria:

* History of psychiatric or personality disorders that may affect the patient's ability to participate
* History of stroke, chronic seizures, or major neurological disorder
* History of clinically significant endocrine, gastrointestinal, cardiovascular, hematological, hepatic, immunological, renal, respiratory, or genitourinary abnormalities or diseases (excluding lipid abnormalities)
* Poorly controlled or recently diagnosed Type 1 or Type 2 diabetes mellitus
* History of neoplastic disease within previous 5 years
* Consumes alcohol or excessive amounts of products that contain caffeine (e.g. cola)
* Has had major surgery, donated and/or received blood within previous 8 weeks
* Participated in another investigational study within previous 4 weeks
* History of significant multiple and/or severe allergies (including latex allergy), or has had an anaphylactic reaction or significant intolerability to prescription or non-prescription drugs or food
* Positive for hepatitis B surface antigen, hepatitis C antibodies or human immunodeficiency virus (HIV)
* Cannot swallow large tablets
* Pregnant or breastfeeding

Ages: 10 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 10 (Actual)
Dates: Start 2012-06; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: MK-0524A-158 was terminated after the Phase 3 study HPS2-THRIVE (MK-0524A-042;NCT00461630) didn't meet its primary endpoint of reduction of major vascular events; there was also a significant increase in some types of non-fatal serious adverse events. MK-0524A-158 was terminated after 10 participants completed Panel A. Panel B was not conducted.
Period: Overall Study
Arm/Group | MK-0524A 1 g/20 mg (Panel A) | MK-0524A 2 g/40 mg (Panel B)
Started | 10 | 0 (Study terminated prior to Panel B being conducted.)
Completed | 10 | 0
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Arm/Group | MK-0524A 1 g/20 mg (Panel A)
Number analyzed (Participants) | 10
Age, Continuous [Mean (Standard Deviation); unit: Years] | 15.4 (0.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 5

OUTCOME MEASURES:

1. Primary Outcome: Plasma Area Under the Concentration Curve From 0 to Infinity (AUC0-∞) of Laropiprant
Time Frame: Predose Day 1 up to 24 hours postdose
Population: The study was terminated during Panel A and the decision was made to not analyze the blood and urine pharmacokinetic samples collected during Panel A; Panel B was not conducted.
Arm/Group | MK-0524A 1 g/20 mg (Panel A) | MK-0524A 2 g/40 mg (Panel B)
Number analyzed (Participants) | 0 | 0

2. Primary Outcome: Plasma Maximum Concentration (Cmax) of Laropiprant
Time Frame: Predose on Day 1 up to 48 hours postdose
Population: as for outcome 1
Arm/Group | MK-0524A 1 g/20 mg (Panel A) | MK-0524A 2 g/40 mg (Panel B)
Number analyzed (Participants) | 0 | 0

3. Primary Outcome: Total Urinary Excretion of Niacin and Niacin Metabolites
Time Frame: Predose on Day 1 up to 72 hours postdose
Population: as for outcome 1
Arm/Group | MK-0524A 1 g/20 mg (Panel A) | MK-0524A 2 g/40 mg (Panel B)
Number analyzed (Participants) | 0 | 0

4. Primary Outcome: Plasma Cmax of Nicotinuric Acid (NUA)
Time Frame: Predose on Day 1 up to 48 hours postdose
Population: as for outcome 1
Arm/Group | MK-0524A 1 g/20 mg (Panel A) | MK-0524A 2 g/40 mg (Panel B)
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: up to 14 days for each panel
Description: MK-0524A-158 was terminated after the Phase 3 study HPS2-THRIVE (MK-0524A-042) didn't meet its primary endpoint of reduction of major vascular events; there was also a significant increase in some types of non-fatal serious adverse events in HPS2-THRIVE. MK-0524A-158 was terminated after 10 participants completed Panel A. Panel B was not conducted.
Arm/Group | MK-0524A 1 g/20 mg (Panel A) | MK-0524A 2 g/40 mg (Panel B)
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/0
Other Adverse Events (participants affected / at risk) | 7/10 | 0/0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MK-0524A 1 g/20 mg (Panel A) (N=10) | MK-0524A 2 g/40 mg (Panel B) (N=0)
Abdominal pain lower (Gastrointestinal disorders) | 1 (1) | 0 (0)
Bruising of arm (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Sprain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Low back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 2 (2) | 0 (0)
Diuresis (Renal and urinary disorders) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Facial flushing (Vascular disorders) | 1 (1) | 0 (0)
Flushing (Vascular disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The SPONSOR must have the opportunity to review all proposed abstracts, manuscripts, or presentations regarding this study 60 days prior to submission for publication/presentation. Any information identified by the SPONSOR as confidential must be deleted prior to submission. SPONSOR review can be expedited to meet publication timelines.